CLINICAL TRIAL: NCT04834999
Title: Validation and Transcultural Adaptation of Instruments Used in a Clinical Trial on Patients With Bipolar Disorder in Rwanda
Brief Title: Validation of Instruments for Clinical Trial on Patients With Bipolar Disorder in Rwanda
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: University of Rwanda (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUUR2020DKRW_4
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2021-04

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of questionnaires in Kinyarwanda — Four questionnaires, three self-report instruments (Medication Adherence Rating Scale, Internalized Stigma of Mental Illness Inventory - 9-item Version and the Mood Disorder Questionnaire) and one clinical interview (the Young Mania Rating Scale)

SUMMARY:
This study evaluates the cultural and linguistic sensitivity and psychometric properties of a set of four adapted measurement instruments essential to determining the efficacy of group-psychoeducation for patients with bipolar disorder in Rwanda, and one screening tool for bipolar disorder. The four well-known instruments are; The Young Mania Rating Scale (YMRS), The Medical Adherence Scale (MARS), The Internalized Stigma of Mental Illness Scale-9 (ISMI-9), and the Mood disorder Questionnaire (MDQ). Each instrument will be culturally adapted and validated using a forward-backward translation, consensus conference, and cognitive interviews.

DETAILED DESCRIPTION:
In the present study, our aim is to translate, culturally adapt and validate four used scales for use in patients with bipolar disorder. The four scales are:

1. The Medical Adherence Scale (MARS), used to assess beliefs and barriers to medication adherence. The scale has 10-items, a total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.
2. Internalized Stigma of Mental Illness Inventory - 9-item Version (ISMI-9) used to assess self-stigma. The scale consists of nine questions evaluated on a four-point Likert scale from 1 (strongly agree) to 4 (strongly disagree). The resulting score should range from 1 to 4. A score ranging between 1.00-2.50: does not report high internalized stigma vs. a score ranging between 2.51-4.00: indicating high internalized stigma
3. The Young Mania Rating Scale (YMRS) is a clinical interview scale to assess the severity of manic states and has 11-items.
4. The Mood Disorder Questionnaire, is a self-reported screening instrument used for identifying persons likely to have bipolar disorder. The instrument comprising a list of 13 hypomanic symptoms.

The translation and adaptation process:

One a nonprofessional translator, bilingual and knowledgeable about mental health care. The second is a translator with no particular knowledge about mental health healthcare. Following the forward translations, a meeting will be held to generate an agreed version. Next, two professional, bilingual, native English speakers back-translated the synthesized version to English. After that, an expert meeting will be held with all translators and five clinicians. Item by item, all versions, and back translations will be discussed to agree on an optimal pre-version for semantic and conceptual equivalence between the original English and the Kinyarwanda version. After that, the tools will be validated among 500 participants.

ELIGIBILITY:
Participants for validation of the YMRS and the MARS:

Inclusion Criteria:

* Patients with a diagnosis of BD type I or II, that meets DSM-IV diagnostic criteria given by a trained psychiatrist

Participants for validation of the ISMI-9:

Inclusion Criteria:

* A diagnosis of mental disorder that meets DSM-IV diagnostic criteria given by a trained psychiatrist

Participants for validation of the MDQ:

Inclusion Criteria:

* Patient with a diagnosis of BD type I or II, or major depression that meets DSM-IV diagnostic criteria given by a trained psychiatrist
* Volunteers with no history or family history of the psychiatric disorder will be recruited as controls.

Exclusion Criteria for all participants:

* Insufficient understanding of Kinyarwanda
* Clinical evidence of substantial cognitive impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a mental illness will be recruited at their scheduled outpatient clinic visit, during which they complete the Kinyarwanda version of the instruments.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Adaption and validation of the Rwandese version of the Mood Disorder Questionnaire for screening for Bipolar Disorder | Ten months
  The study aims to adapt and validate the Mood Disorder Questionnaire to improve the detection of bipolar disorder in Rwanda
Adaption and validation of the Rwandese version of the Medication Adherence Rating Scale (MARS). | Ten months
  The study aims to adapt and validate the Medication Adherence Rating Scale (MARS) and to access the medical adherence
Adaption and validation of the Rwandese version of The Internalized Stigma of Mental Illness Scale-9 (ISMI-9) | Ten months
  The study aims to adapt and validate The Internalized Stigma of Mental Illness Scale-9 (ISMI-9) to measure the overall self-stigma of mental illness among persons with psychiatric disorders in Rwanda.
Adaption and validation of the Rwandese version of the Young Mania Rating Scale | Ten months
  The study aims to adapt and validate the Young Mania Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Per Kallestrup, Prof., Study Chair — University of Aarhus
Locations (1):
- The University Teaching Hospital of Kigali (CHUK) and Ndera Hospital, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No